CLINICAL TRIAL: NCT03546595
Title: Effect of Auricular Points Acupressure for Overweight/Obese Women With Polycystic Ovary Syndrome.
Brief Title: Auricular Acupressure (AA) For Insulin Resistance in Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yan Li, Associate chief physician, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AA for IR-PCOS
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
Keywords: Polycystic Ovary Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupoints acupressure (Experimental)
  Interventions: Other: Auricular acupoints acupressure
- Sham auricular acupoints acupressure (Sham Comparator)
  Interventions: Other: Sham auricular acupoints acupressure

INTERVENTIONS:
Other: Auricular acupoints acupressure — The magnetic beads were taped to the auricular acupressure points, by the same acupuncture specialist on one ear approximately after skin sterilization, and the subjects were asked to massage the points for 5 minutes, 30 minutes before three meals and sleep.The magnetic beads were left in situ, but replaced with new ones once every week in the other ear.
  Arms: Auricular acupoints acupressure
Other: Sham auricular acupoints acupressure — The magnetic beads were taped to the auricular acupressure points, by the same acupuncture specialist on one ear approximately after skin sterilization, and the subjects were not asked to massage the points.The magnetic beads were left in situ, but replaced with new ones once every week in the other ear.
  Arms: Sham auricular acupoints acupressure

SUMMARY:
The present trial is a pilot study to investigate the effect of auricular acupressure on insulin resistance in women with PCOS.A total of 100 subjects will be enrolled into this study and will be randomized into two groups.

Auricular acupressure or sham auricular acupressure will be treated for three months. The primary outcome is the whole body insulin action assessed with HOMA-IR.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 15 and 40 years.
* Diagnosis of PCOS according to the modified Rotterdam criteria.
* 2 years after menarche.
* Body mass index (BMI) equal to or greater than 23 kg/m2.
* IR is defined by the homeostaticmodel assessment (HOMA-IR: (fasting insulin (μU/mL)×fasting glucose (mmol/L))/22.5). A value ≥2.14 will be considered to be indicative of IR.
* With no desire of children within 3 months.

Exclusion Criteria:

* Administration of other medications known to affect reproductive function or metabolism within the past three months, including oral contraceptives, Gonadotropin-releasing hormone (GnRH) agonists and antagonists, anti androgens, gonadotropins, anti-obesity drugs, Chinese herbal medicines, anti diabetic drugs such as metformin and thiazolidinediones, somatostatin, diazoxide, and calcium channel blockers.
* Patients with other endocrine disorders including 21-hydroxylase deficiency, hyperprolactinemia, uncorrected thyroid disease, suspected Cushing's syndrome.
* Patients with known severe organ dysfunction or mental illness.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Homeostasis model assessment-insulin resistance (HOMA-IR) | 3 month
  HOMA-IR was calculated as [Plasma glucose (GLU,mmol/L)* serum insulin (mIU/L)] / 22.5.

SECONDARY OUTCOMES:
Testosterone(T) | 3 month
Androstadienedione (AND) | 3 month
Sex hormone-binding globulin (SHBG) | 3 month
Dehydroepiandrosterone sulfate (DHEAS) | 3 month
Follicle stimulating hormone (FSH) | 3 month
Luteinizing hormone (LH) | 3 month
Estradiol (E2) | 3 month
Weight | 3 month
Waist/hip circumference | 3 month
BMI | 3 month
FG score | 3 month
Acne | 3 month
Short-Form Health Survey (SF-36) | 3 month
The Chinese Quality of Life questionnaire (ChQoL) | 3 month
Health-related quality of life questionnaire for polycystic ovary syndrome (PCOSQ) | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Hou L, Wang Y, Xie L, Zhang M, Pan Z, Li Y, Ding Y, Sun M, Qu Y, Liu S. Auricular points acupressure for insulin resistance in overweight/obese women with polycystic ovary syndrome: protocol for a randomised controlled pilot trial. BMJ Open. 2019 May 28;9(5):e027498. doi: 10.1136/bmjopen-2018-027498. PMID 31142530